CLINICAL TRIAL: NCT05925660
Title: Mucorales PCR Screening in At-risk Hematology Patients
Acronym: MUCOPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: AZ Sint-Jan AV (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: S67347; IN-EU-131-6808 (Other Grant/Funding Number: Gilead Sciences); S-number CTC UZ Leuven (Other: S67347)
Record Dates: First submitted 2023-06-15; First posted 2023-06-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-06

CONDITIONS: Mucormycosis
Keywords: Invasive Mycosis; Neutropenia; Leukemia; Stem Cell Transplant Complications; Invasive Mucormycosis
MeSH Terms: conditions — Mucormycosis; Invasive Fungal Infections; Neutropenia; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Mucorales PCR (MucorGenius, PathoNostics, Maastricht, The Netherlands) — Mucorales PCR screening twice weekly during hospitalisation

SUMMARY:
Patients with leukemia are treated with intensive chemotherapy and often have to undergo a stem cell transplantation which makes their immune system extremely vulnerable. This puts them at risk for invasive fungal infections, of which invasive mucormycosis (IM) is one of the most dangerous ones. Treatment of IM is complex and mortality rates are still extremely high, ranging from 40% to 80% and sometimes even higher if the central nervous system is involved. Mucormycosis requires immediate intervention due to the rapidly progressive and destructive nature of the infection. But the diagnosis is often made too late…

Better survival can be achieved with a faster diagnosis. A new test has recently been developed for detection of Mucorales DNA by PCR. The polymerase chain reaction (PCR) is a method that allows to quickly make millions of copies of, for example, Mucorales DNA in order to detect it in the blood at an early stage. Because blood can easily be obtained, without an additional burden on the patient, the test could be interesting for screening for these infections, which then offers the opportunity to start an adequate treatment more quickly.

However, the test is now only performed if there is a clinical suspicion of IM. But at that point, precious time has already been lost, and often the patient can no longer be cured. In this study the utility of the Mucorales PCR as a possible screening test in at-risk patients is assessed. The participants, hospitalised patients with leukemia, will be screened twice weekly with a Mucorales PCR test during their most vulnerable period. If the study shows that the test helps in diagnosing IM faster, this could have an important impact on the treatment and survival of these at-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Underlying disease:

  * Start of remission induction chemotherapy for acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) that is newly diagnosed or in first relapse after hematological remission lasting for a minimum duration of 6 months; OR
  * Start of myeloablative conditioning regimen to prepare for a first allogeneic hematopoietic cell transplantation (HCT).
* Expected prolonged neutropenia (ANC< 0.5 x 109 /L for ≥ 7 days).
* Planned hospital admission for the duration of the neutropenic phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of a positive Mucorales PCR screening test | 3 months

SECONDARY OUTCOMES:
Incidence of invasive mucormycosis | 3 months
Incidence of invasive aspergillosis and invasive mucormycosis coinfections | 3 months
Number of days antifungal therapy was given (amphotericin B, azoles) | 3 months
Was antifungal therapy started based on Mucorales PCR result? Y/N | 3 months
Was antifungal therapy stopped based on Mucorales PCR result? Y/N | 3 months
Outcome of patients with a positive Mucorales PCR versus these without: death or survival at 3 months | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No